CLINICAL TRIAL: NCT02836678
Title: Bone Changes in Atrophic Maxilla Treated by Split-crest Technique and Dental Implants With Platelet Rich Fibrin and Nanobone® Versus Platelet Rich Fibrin Alone; Randomized Controlled Trial
Brief Title: Bone Changes in Atrophic Maxilla Treated by Split-crest Technique
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Wadie Anis, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-2016-03-150
Record Dates: First submitted 2016-07-11; First posted 2016-07-19 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Atrophy; Edentulous Ridge
MeSH Terms: conditions — Atrophy | interventions — NanoBone; Prolactin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): Ridge splitting, immediate implantand PRF.
  Interventions: Biological: Ridge splitting, immediate implantand PRF.
- Test group (Experimental): Ridge splitting, immediate implant, Nanobone with PRF.
  Interventions: Biological: Ridge splitting, immediate implant, Nanobone with PRF.

INTERVENTIONS:
Biological: Ridge splitting, immediate implant, Nanobone with PRF. — * Dental implant (is a surgical component that interfaces with the bone of the jaw or skull to support a dental prosthesis).
  * Alloplast bone graft material (Nanobone)
  * PRF platelet rich fibrin. (second-generation Platelet rich plasma where autologous platelets and leucocytes are present in a complex fibrin matrix to accelerate the healing of soft and hard tissue).
  Arms: Test group
Biological: Ridge splitting, immediate implantand PRF. — * Dental implant (is a surgical component that interfaces with the bone of the jaw or skull to support a dental prosthesis).
  * PRF platelet rich fibrin. (second-generation Platelet rich plasma where autologous platelets and leucocytes are present in a complex fibrin matrix to accelerate the healing of soft and hard tissue).
  Arms: Control group

SUMMARY:
The effect of adding Nanobone on horizontal bone gain in ridge splitting.

DETAILED DESCRIPTION:
In cases of a very narrow ridge, One of the augmentation protocols is alveolar ridge-splitting techniques (RST) or alveolar ridge expansion techniques with simultaneous implant insertion. The piezoelectric surgical devices implemented for conducting bone osteotomy through the use of micrometric ultrasonic vibrations have been widely used in recent years in maxillofacial surgery. Its biggest advantages are that it allows for cutting with micrometric sensitivity while cutting hard tissues, it offers a clear vision of the surgical site due to its cavitation effect, it does not cause any damage to the soft tissues while performing these cuts, and that the bone tissue heals more quickly and seamlessly, after the cuts made by piezosurgery device. The fully synthetic bone substitute, NanoBone® (Artoss, Rostock, Germany), which will be applied in this clinical study, is basically a nanocrystalline hydroxyapatite embedded in a silica gel matrix, achieved by means of specific sol-gel techniques. Features such as interconnecting pores on the nanoscale, the open SiOH or SiO groups of polysilicic acid, its large internal surface, and the high porosity of this biomaterial are all related to the calcification processes observed within the implantation bed. While the HA component is responsible for NanoBone osteoconductive properties, the silica component is believed to induce connective tissue formation, osteoblast proliferation, bone matrix mineralization, and calcification, thus combining osteoconductive and osteoinductive properties. This phenomenon is associated with the rearrangement of the silica matrix, which could be observed in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70.
* Patients with an edentulous site in maxilla.
* Ridge width of <6mm at the edentulous site.
* Ridge height of >9mm at the edentulous site.
* Patients who are compliant to oral hygiene measures for 4 weeks.
* Patient consent approval and signing.

Exclusion Criteria:

* Smokers.
* Systemic disease that contraindicates implant placement or surgical procedures.
* No or poor patient's compliance.
* History of radio or chemo-therapy.
* Psychological problems.
* Pathology at the site of intervention.
* Pregnancy.
* Insufficient crown height space or mesio-distal dimension that contradict the placement of a dental implant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone gain in millimeters | 5 month
  using Cone beam computed tomography

SECONDARY OUTCOMES:
Post-operative pain Using Numerical rating scale | 2 weeks
Post-operative swelling Using Descriptive 4-point scale of swelling | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amr Zahran, Professor, Study Chair — Professor of Oral Medicine, Periodontology and Oral Diagnosis; Ahmed Reda, Lecturer, Study Director — Lecturer of Oral Medicine, Periodontology, and Oral Diagnosis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gerber, T., Holzhüter, G., Knoblich, B., Dörfling, P., Bienengräber, V., & Henkel, K. O. (2000). Development of bioactive sol-gel material template for in vitro and in vivo synthesis of bone material. Journal of Sol-Gel Science and Technology, 19(1-3), 441-445. http://doi.org/10.1023/A:10087995
- [Background] Porter AE, Patel N, Skepper JN, Best SM, Bonfield W. Effect of sintered silicate-substituted hydroxyapatite on remodelling processes at the bone-implant interface. Biomaterials. 2004 Jul;25(16):3303-14. doi: 10.1016/j.biomaterials.2003.10.006. PMID 14980425
- [Derived] Anis M, Abdelrahman AR, Attia R, Zahran A. Tomographic assessment of bone changes in atrophic maxilla treated by split-crest technique and dental implants with platelet-rich fibrin and NanoBone(R) versus platelet-rich fibrin alone: Randomized controlled trial. BMC Oral Health. 2024 Jun 14;24(1):691. doi: 10.1186/s12903-024-04420-5. PMID 38877464